CLINICAL TRIAL: NCT05209789
Title: HUGS : Early Intervention to Protect the Mother-Child Relationship After Postpartum Depression: A Randomized Comparative Trial of the Cognitive Behavioral Therapy Program
Brief Title: Early Intervention to Protect the Mother-Child Relationship After Postpartum Depression
Acronym: HUGS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC31/21/0166
Record Dates: First submitted 2022-01-11; First posted 2022-01-27 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Post Partum Depression
Keywords: Mother-baby interaction; Group therapy; Cognitive behavioral therapy; mother-infant relationship
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Multicenter, interregional, comparative, prospective therapeutic study in 2 parallel groups (1: 1), superiority, randomized, blinded for the evaluation of the primary endpoint.
Who Masked: Participant
Masking Description: group attribution blinded to evaluators for the evaluation of the primary endpoint via video tapes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HUGS therapy (Experimental): A structured group intervention that aims to observe mother's behavior and responses with her baby, promote mother-baby interaction through play, and provide tools for positive interaction. This therapy involves cognitive and behavioral work. Therapists observe the mother-baby duo and share their observations from a perspective of encouragement and support. A playful and non-judgmental interaction is cultivated within the group. The main objective is to change the negative trajectory of mother-child interactions through tools from cognitive-behavioral therapies as well as using knowledge about child development.
  Interventions: Behavioral: HUGS
- Playtime (Active Comparator): The participants assigned to the control group will also be in the presence of two therapists, allowing to reproduce the framework of the HUGS therapy. The difference will be the lack of direct therapeutic intervention from the therapists, but only classic psychoeducational guidance. The mothers are offered a time to play with their baby as well as the opportunity to discuss and share their experiences with other mothers, which is generally seen as supportive by them.
  Interventions: Behavioral: Playtime

INTERVENTIONS:
Behavioral: HUGS — Group therapy with the participation of two therapist positively encouraging mother-baby interactions in a non-judgmental manner
  Arms: HUGS therapy
Behavioral: Playtime — Very little intervention from the therapists
  Arms: Playtime

SUMMARY:
Postpartum depression (PPD) may impair the mother-infant relationship and lead to both short and long-term suboptimal development of the baby. This study aims to evaluate the effectiveness of a targeted intervention (HUGS: Happiness Understanding Giving and Sharing) for enhancing the mother-infant relationship.

DETAILED DESCRIPTION:
Post-partum depression (PPD) is the most common psychological pathology following childbirth and affects 12% of women in France. This pathology may impair the mother-infant relationship and lead to suboptimal development of the baby in the short and long-term. The prevalence of early interaction disorders is estimated at 73% among women suffering from PPD. Although treatments for PDD are effective, the mother-infant interaction remains impaired, as well as the short, medium and long-term development of the child. It is therefore essential to develop at a very early stage an intervention specifically targeting the mother-infant interaction, and to integrate this care into the general care given to mothers suffering from PPD.

A short cognitive-behavioural therapy intervention focused on improving the quality of the mother-infant relationship (the HUGS program: Happiness, Understanding, Giving and Sharing) has been created and validated by Prof. Jeannette Milgrom's Australian team. The objective of our study is to evaluate the effectiveness of the HUGS programme compared to a Playtime control group using a randomised controlled trial in a population of women suffering from PPD and being cared for in 7 French maternity hospitals. The comparison will be made 6 months after intervention initiation using "Factor 1: Mother Positive Affective Involvement and Verbalization" of the PCERA (Parent-Child Early Relational Assessment) mother-child interaction evaluation scale.

ELIGIBILITY:
Inclusion criteria regarding the mother:

* Person affiliated or beneficiary of a social security plan;
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research);
* Woman who gave birth in one of the maternity hospitals participating in the study;
* Diagnosis of postpartum depression made by the perinatal psychiatry team according to the clinical criteria of the DSM-5;
* Time to onset of depressive symptoms within the first 12 months after childbirth;
* Treatment for postpartum depression that started at least 8 weeks ago with improved mood as assessed by the psychiatrist.

Inclusion criteria for the baby:

* Baby aged less than 1 year at inclusion;
* Twins will be able to participate in the study and benefit from the interventions;

Non-inclusion criteria concerning the mother:

* Uncontrolled substance use disorder;
* Presence of suicidal ideas at inclusion;
* Manic episode of a bipolar disease
* Psychiatric pathology decompensated upon inclusion and corresponding to the following list: Schizophrenic disorder, Schizoaffective disorder, Mood disorders with psychotic symptoms;
* Non French speaker.

Non-inclusion criteria for the baby:

- Baby hospitalized or having sustained medical care upon inclusion in the context of a somatic pathology.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Mothers
Enrollment: 104 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mother-infant interaction | 6 months after the end of the intervention
  The primary endpoint will be the score of factor 1 ("positive affective commitment of the mother as well as her verbalization skills with her baby") of the mother-baby interaction assessment scale The Parent-Child Early Relational Assessment ( PCERA) between the two study groups : HUGS and Playtime.
  PCERA factor 1 will be measured by analysis of video footage of each mother-baby duo by two independent blind assessors from allocation groups.The score taken into account will be the consensus score between the two evaluators.

SECONDARY OUTCOMES:
Mothers' stress | Right before the intervention (Baseline)
  Parental Stress Index (PSI-3) measured on both groups. This index is categorised in various items (stressors), each including a Likert style index from 1 to 5. The PSI-3 sums up all the items into a score : a high score representing a high stress for the parent.
Mothers' stress | Right at the end of the intervention : 28 days after the start of the study
  Parental Stress Index (PSI-3) measured on both groups. This index is categorised in various items (stressors), each including a Likert style index from 1 to 5. The PSI-3 sums up all the items into a score : a high score representing a high stress for the parent.
Mothers' stress | 6 months after the end of the intervention
  Parental Stress Index (PSI-3) measured on both groups. This index is categorised in various items (stressors), each including a Likert style index from 1 to 5. The PSI-3 sums up all the items into a score : a high score representing a high stress for the parent.

OTHER OUTCOMES:
Socio-economic analysis | 6 months after the end of the intervention
  the efficiency of the HUGS program compared to usual care, by means of a cost-utility analysis: Costs of support from the point of view of the community and QALYs in order to calculate a differential cost-utility ratio (collected using the EUROQOL EQ-5D-5L scale).

CONTACTS AND LOCATIONS:
Overall Officials: Carole GENTILLEAU, MD, Principal Investigator — University Hospital, Toulouse
Locations (7):
- France (7):
  - Bordeaux Public Hospital, Bordeaux
  - Havre Public Hospital Maternity, Le Havre
  - Reims Public Hospital Maternity, Reims
  - Rouen Public Hospital Maternity, Rouen
  - Toulouse Child Guidance, Toulouse
  - Toulouse Joseph Ducuing Maternity, Toulouse
  - Toulouse Public Hospital Maternity, Toulouse